CLINICAL TRIAL: NCT06679387
Title: "The Effect of Memantine on the Prevention and Amelioration of Paclitaxel-induced Toxicity in Breast Cancer Patients"
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mahmoud Mustafa Mahmoud Gharib, Assistant lecturer at Pharmacy Practice & Clinical Pharmacy Department, Future University in Egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 45
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Paclitaxel-induced Toxicity; Breast Cancer patients; Memantine; Neurotoxicity Prevention or treatment
MeSH Terms: interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Forty patients who will receive memantine 20 mg once daily in addition to weekly 80 mg/m2 of paclitaxel for 12 weeks.
  Interventions: Drug: Memantine-HCl
- Control arm (Placebo Comparator): Forty patients who will receive placebo once daily in addition to weekly 80 mg/m2 of paclitaxel for 12 weeks.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Memantine-HCl — Memantine hydrochloride 20 mg once daily for 12 weeks.
  Other Names: Memantine 20 mg
  Arms: Treatment arm
Drug: Placebo Oral Tablet — A once daily matched tablet of placebo for 12 weeks
  Other Names: Placebo comparator
  Arms: Control arm

SUMMARY:
Cancer is currently a leading cause of morbidity and mortality worldwide. Chemotherapeutic agents, despite being effective in arresting the progression of cancer by targeting and eliminating rapidly dividing cancer cells, are associated with various adverse effects. Chemotherapy-induced peripheral neuropathy (CIPN) is a serious clinical adverse effect of certain chemotherapeutic agents. For many patients, CIPN symptoms could be severe, disabling, and significantly impairing the activities of daily living (ADL) and diminishing the quality of life (QoL). Paclitaxel-induced peripheral neuropathy may affect up to 97% of paclitaxel-treated patients and become chronic in more than 60% of cases. The initial symptoms of paclitaxel-induced peripheral neuropathy (PIPN) include numbness, tingling, and allodynia (painful sensations in response to normally non-painful stimuli) that can be manifested in the patient's fingers and toes within 24-72 h post-injection. These symptoms may later progress to affect the patient's lower leg and wrists in a "glove and stocking" pattern. Symptoms typically begin distally and continue proximally as the situation worsens. Memantine is a non-competitive NMDA receptor antagonist that inhibits the prolonged influx of Ca2+, responsible for neuronal excitotoxicity while maintaining the physiological NMDA receptor's function and avoiding psychotropic adverse events. Although memantine has been the main treatment option for moderate and severe Alzheimer's disease in the last two decades, numerous studies have investigated its other potential uses. Some studies showed that memantine diminished chronic pain in complex regional pain syndrome, phantom limb pain, and fibromyalgia. Most in vivo and in vitro studies attributed the neuroprotective effects of memantine to the blockade of NMDA receptors on neurons as well as inhibition of microglia activation with subsequent reduction of pro-inflammatory mediators' production such as extracellular superoxide anion, intracellular ROS, nitric oxide, prostaglandin E2, and TNF-α, and stimulation of neurotrophic factor release from astroglia.

DETAILED DESCRIPTION:
Up till now, no treatment options are available for prevention of PIPN. Several options have been investigated for treatment of CIPN with only duloxetine had proven benefits. Additional investigations are needed to develop preventive and ameliorative therapy of PIPN.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old).
* Patients with confirmed diagnosis of non-metastatic breast cancer planned to receive weekly adjuvant/neo-adjuvant paclitaxel.
* Patients with Eastern Cooperative Oncology Group (ECOG) performance (Oken et al., 1982) status of 0-2.

Exclusion Criteria:

* Patients with pre-existing neuropathic conditions.
* Patients with diabetes mellitus.
* Patients with a history of seizure disorder.
* Patients with renal impairment (creatinine clearance less than 60 ml/min), or hepatic impairment (defined as ALT an AST > 3 times upper limits of normal)
* Patients with inadequate bone marrow functions (defined as absolute neutrophilic count less than 1,500/mm3 or platelets count less than 100,000/mm3).
* Concomitant use of vitamin B1, B6, B9, or B12.
* Patients receiving medications that possibly induce peripheral neuropathy including amiodarone, colchicine, metronidazole, antimycobacterials, and nucleoside reverse transcriptase inhibitors, and phenytoin (Jones et al., 2020).
* Patients receiving gabapentinoids, antidepressants, or opioids.
* Pregnancy or lactation.
* History of hypersensitivity to memantine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and grading of paclitaxel induced peripheral neuropathy (PIPN) | Weekly for 12 weeks.
  Patients will be subjected to neurological examination every cycle to identify the presence and severity of PIPN. Grading of PIPN will be determined using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5 published in November 2017 (NCI, 2017). The NCI-CTCAE grades the adverse events based on their severity on a 5-point scale where "Grade 1" is defined as: Mild or asymptomatic symptoms requiring clinical or diagnostic observations only; Intervention not indicated. "Grade 2": Moderate symptoms limiting age-appropriate ADL; minimal, local or noninvasive intervention is indicated. "Grade 3": Severe symptoms or medically significant but not life-threatening that are disabling or limiting self-care in ADL; hospitalization or prolongation of hospitalization is indicated. "Grade 4": Life threatening consequences; urgent or emergent intervention is needed. "Grade 5": Death related to adverse event. The primary outcome will be the difference i

SECONDARY OUTCOMES:
Pain severity | Weekly for 12 weeks.
  Pain severity will be quantified using the Brief Pain Inventory Short Form (BPI-SF) (Cleeland and Ryan, 1994). It is widely used in both research and clinical settings. Patients will be asked to rate their pain on a numerical scale every cycle. Each scale is presented as a row of equidistant numbers from zero to ten, where zero indicates "no pain" and ten indicates "pain as bad as you can imagine".
Patients' QoL | baseline, at 6 weeks, and 12 weeks.
  Patients' QoL will be assessed through The Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity subscale (FACT/GOG-Ntx) questionnaire. The Ntx subscale is a reliable and valid instrument for assessing the impact of neuropathy on QoL that demonstrates sensitivity to meaningful clinical distinctions and change over time.
  It is an eleven-item subscale that evaluates sensory neuropathy, motor neuropathy, hearing neuropathy, and dysfunction associated with CIPN for the previous 7 days. Each question in the Ntx subscale is represented by a Likert scale ranging from zero to four, where zero represents "not at all" and four represents "very much". The Ntx subscale generates a total score that is obtained by the summation of the composing question's scores. The total score ranges from 0 to 44 with higher scores indicating more severe neurotoxicity and worse QoL. The FACT/GOG-Ntx subscale will be evaluated at baseline, at 6 weeks, and 12 weeks.
Serum levels of nerve growth factor (NGF) | Baseline and at 12 weeks.
  Nerve growth factor, one of major neurotrophins, is known to regulate the growth, maintenance, and survival of neurons. Clinical evidence supports that depletion of NGF occurs during the development of CIPN. In cancer patients receiving taxanes, serum levels of NGF levels were shown to decrease after four to six cycles and decline was associated with the severity of PIPN. For the determination of serum levels of NGF, a blood sample of 4 ml will be collected from every patient.
Severity of depressive symptoms | Baseline, at 6 weeks, and 12 weeks.
  The effect of memantine on depressive symptoms will be assessed through the nine-items Patient Health Questionnaire (PHQ-9). It is an easy-to-use self-administered questionnaire that reflects each of the nine criteria that the diagnosis of depression is based on according to the Diagnostic and Statistical Manual of Mental Disorders version V (DSM-V) criteria. The score for each question ranges from 0-3, as "0" (not at all) to "3" (nearly every day). The total score is obtained by adding up the individual items' scores. Scores range from 0 to 27 with scores from 0-4 indicating minimal depressive symptoms, 5-9: Mild, 10-14: Moderate, 15-19: Moderately severe, 20-27: Severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folch J, Busquets O, Ettcheto M, Sanchez-Lopez E, Castro-Torres RD, Verdaguer E, Garcia ML, Olloquequi J, Casadesus G, Beas-Zarate C, Pelegri C, Vilaplana J, Auladell C, Camins A. Memantine for the Treatment of Dementia: A Review on its Current and Future Applications. J Alzheimers Dis. 2018;62(3):1223-1240. doi: 10.3233/JAD-170672. PMID 29254093
- [Background] Argyriou AA, Koltzenburg M, Polychronopoulos P, Papapetropoulos S, Kalofonos HP. Peripheral nerve damage associated with administration of taxanes in patients with cancer. Crit Rev Oncol Hematol. 2008 Jun;66(3):218-28. doi: 10.1016/j.critrevonc.2008.01.008. Epub 2008 Mar 7. PMID 18329278